CLINICAL TRIAL: NCT03214718
Title: Effect of Tyrosine Kinase Inhibitors on Myeloid Derived Suppressor Cells in Chronic Myeloid Leukemia Patients
Brief Title: Myeloid Derived Suppressor Cells and Chronic Myeloid Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yomna Refaat Mahboub, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDCSCML
Record Dates: First submitted 2017-07-03; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Chronic Myeloid Leukemia Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CML patients treated with imatinib 400 mg/day (Experimental): Measurement of the level of myeloid derived suppressor cells (MDSCs) by flowctytometry for each newly diagnosed chronic phase chronic myeloid leukemia (CML) patients treated with imatinib 400 mg/day before starting treatment and every 3 months till one year and correlate between it and level of BCR-ABL gene level and the sokal score of the patients and deep molecular response of the patients after one year .
  Interventions: Diagnostic Test: Measurement level of myeloid derived suppressor cells in CML patients treated with imatinibe 400 mg/day
- CML patients treated with nilotinib 600 mg/day (Active Comparator): Measurement of the level of myeloid derived suppressor cells (MDSCs) for each newly diagnosed chronic phase chronic myeloid leukemia ( CML) patients treated with nilotinib 600 mg/day before starting treatment and every 3 months till one year and correlate between it and level of BCR-ABL gene, the sokal score and deep molecular response of the patients after one year .
  Interventions: Diagnostic Test: Measurement level of myeloid derived suppressor cells in CML patients treated with nilotinib 600 mg/day

INTERVENTIONS:
Diagnostic Test: Measurement level of myeloid derived suppressor cells in CML patients treated with imatinibe 400 mg/day — For each patient these investigation will be done:
  - Complete blood count,bone marrow aspirate and bone marrow biopsy Measure BCR-ABL GENE Level by FISH at diagnosis and every 3 months till one year .
  Measurement Level of myeloid derived suppressor cells both granulocytic and monocytic cells by flowcytometry .
  Arms: CML patients treated with imatinib 400 mg/day
Diagnostic Test: Measurement level of myeloid derived suppressor cells in CML patients treated with nilotinib 600 mg/day — For each patient these investigation will be done:
  - Complete blood count,bone marrow aspirate and bone marrow biopsy Measure BCR-ABL GENE Level by FISH at diagnosis and every 3 months till one year .
  Measurement Level of myeloid derived suppressor cells both granulocytic and monocytic cells by flowcytometry .
  Arms: CML patients treated with nilotinib 600 mg/day

SUMMARY:
The suppression of the immune system creates a permissive environment for development and progression of cancer. One population of immunosuppressive cells that have become the focus of intense study is myeloid derived suppressor cells , immature myeloid cells able to induce immune-escape, angiogenesis, and tumor progression. Two different subpopulations have been identified and studied: granulocytic and monocytic myeloid derived suppressor cells with a different immunophenotype and immunosuppressive properties

DETAILED DESCRIPTION:
Myeloid-derived suppressor cells utilize different mechanisms to block both innate and adaptive arms of anti-tumour immunity, mostly through inhibition of T cell activation and expansion . Human monocytic myeloid derived suppressor cells are mostly identified as CD14+ cells with negative or low expression of HLADR. And also express high levels of CD11b and CD33 antigen . Human granulocytic myeloid derived suppressor cells are usually defined as CD66b+ CD11b+ CD15+ HLADR- cells and display an intermediate expression of CD33 and a variable expression of CD11b, depending on their maturation stage .

Chronic myeloid leukemia (CML) is a hematological cancer, characterized by a reciprocal chromosomal translocation between chromosomes 9 and 22 [t(9;22)], producing the Bcr-Abl oncogene. Tyrosine kinase inhibitors represent the standard of care for CML patients and exert a dual mode of action: direct oncokinase inhibition and restoration of effector-mediated immune surveillance, which is rendered dysfunctional in CML patients at diagnosis, prior to TKI therapy. TKIs such as imatinib, and more potent second-generation nilotinib and dasatinib induce a high rate of deep molecular response (DMR, BCR-ABL1 ≤ 0.01%) in CML patients. As a result, the more recent goal of therapy in CML treatment is to induce a durable deep molecular response as a prelude to successful treatment-free remission .

Accumulation of both Gr-MDSCs and Mo-MDSCs cells has been found in the peripheral blood of chronic myeloid leukemia (CML) patients. They are part of the tumor clone showing BCR/ABL expression.

BCR-ABL tyrosine kinase inhibitors (TKI) are able to induce remission in CML patients but not to eliminate leukemia stem cells , which can regenerate leukemia on drug discontinuation .

Unfortunately, molecular relapse is observed after cessation of tyrosine kinase inhibitors in 61-66% of CML patients, previously in complete molecular response (presumably due to the reactivation of dormant CML LSCs that are resistant to TKI-induced leukemic cell ablation. Thus, current research efforts aim to develop additional therapies to target these TKI-refractory CML LSCs .

With the aim of increasing cure rates and make it possible for patients to discontinue treatment, TKI therapies are currently evaluated in combination with immune modulators .

ELIGIBILITY:
Inclusion Criteria:

* All newly diagnosed chronic phase CML patients during one year in Assiut university hospital.

Exclusion Criteria:

* Preivously diagnosed CML patients .
* Other myeloproliferative disorders .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-08-05 (Estimated); Primary Completion 2019-08-05 (Estimated); Study Completion 2019-08-05 (Estimated)

PRIMARY OUTCOMES:
The effect of the different types of tyrosine kinase inhibitors (TKI) ( imatinib and nilotinib) therapy on MDSC and possible correlation with clinical response. | one years
  measuring response rate of patients on TKIs whether imatinib 400mg/ day or nilotinib 600 mg / day by assessment of level of BCR-ABL gene level measured by FISH in %every 3 months till one year. and correlate between this level and between level of MDSCs measured in % ,.Granulocytic MDSCs (G-MDSCs) were identified as CD11b+CD33+CD14-HLADR- cells, while the monocytic MDSCs (M-MDSCs) as CD14+HLADR by cytofluorimetric analysis also measured every 3 months till one year,and detect if there is decline in level of MDSCs after one year of TKIs therapy.

SECONDARY OUTCOMES:
Relation between the level of (MDSC) and clinical feature and sokal score of CML patients .. | one year
  correlate between MDSCs and clinical features of CML patients as spleen size measured in centimeters, haemoglobin level measured in gram/dl, sokal score of the patients exp (0.0116 x (age [years] - 43.4)) + (0.0345 x (spleen size [cm] - 7.51) + (0.188 x ((platelets [109/L]/700)^2 - 0.563)) + (0.0887 x (blasts [%] - 2.10)).
  low-risk (Sokal score < 0.8), intermediate-risk (Sokal score 0.8 - 1.2) and high-risk (> 1.2 ) .

REFERENCES:
- [Background] Brandau S, Moses K, Lang S. The kinship of neutrophils and granulocytic myeloid-derived suppressor cells in cancer: cousins, siblings or twins? Semin Cancer Biol. 2013 Jun;23(3):171-82. doi: 10.1016/j.semcancer.2013.02.007. Epub 2013 Feb 28. PMID 23459190
- [Background] Giallongo C, Parrinello N, Tibullo D, La Cava P, Romano A, Chiarenza A, Barbagallo I, Palumbo GA, Stagno F, Vigneri P, Di Raimondo F. Myeloid derived suppressor cells (MDSCs) are increased and exert immunosuppressive activity together with polymorphonuclear leukocytes (PMNs) in chronic myeloid leukemia patients. PLoS One. 2014 Jul 11;9(7):e101848. doi: 10.1371/journal.pone.0101848. eCollection 2014. PMID 25014230
- [Background] Christiansson L, Soderlund S, Mangsbo S, Hjorth-Hansen H, Hoglund M, Markevarn B, Richter J, Stenke L, Mustjoki S, Loskog A, Olsson-Stromberg U. The tyrosine kinase inhibitors imatinib and dasatinib reduce myeloid suppressor cells and release effector lymphocyte responses. Mol Cancer Ther. 2015 May;14(5):1181-91. doi: 10.1158/1535-7163.MCT-14-0849. Epub 2015 Mar 11. PMID 25761894
- [Background] Xishan Z, Guangyu A, Yuguang S, Hongmei Z. The research on the immuno-modulatory defect of mesenchymal stem cell from Chronic Myeloid Leukemia patients. J Exp Clin Cancer Res. 2011 May 2;30(1):47. doi: 10.1186/1756-9966-30-47. PMID 21535879